CLINICAL TRIAL: NCT04134442
Title: Improving Pain Management After Total Shoulder Replacement Using Bupivacaine Liposome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: A new large meta-analysis was published. The results showed the likelihood that liposomal bupivacaine and nerve blocks no longer offer significant contribution. Decision was made to terminate the study.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Alexander Chan, Principle-Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H00016941
Record Dates: First submitted 2019-10-02; First posted 2019-10-22 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis of the Shoulder; Shoulder Pain; Pain, Postoperative
Keywords: Exparel; Bupivacaine Liposome; Total Shoulder Replacement; Pain Management
MeSH Terms: conditions — Shoulder Pain; Pain, Postoperative; Agnosia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine Liposome (Experimental): 1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, age, or current therapy as currently determined by APS anesthesiologist).
  2. Pre-operative ultrasound guided ISNB with a 20ml mixture consisting of 10ml of 0.5% bupivacaine with epinephrine 1:200,000, and 10ml of BL 1.33%
  Interventions: Drug: Bupivacaine Liposome Injection
- Standard therapy (Active Comparator): 1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, or age as currently determined by acute pain service (APS) anesthesiologist).
  2. Preoperative, ultrasound guided ISNB with a bupivacaine mixture: 20ml 0.5% bupivacaine and epinephrine 1:200,000.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection — 1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, age, or current therapy as currently determined by APS anesthesiologist)
  2. Pre-operative ultrasound guided ISNB with a 20ml mixture consisting of 10ml of 0.5% bupivacaine with epinephrine 1:200,000, and 10ml of BL 1.33%
  Other Names: Standard Therapy and Bupivacaine Liposome 10ml 1.33%
  Arms: Bupivacaine Liposome
Other: Standard Therapy — 1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, or age as currently determined by acute pain service (APS) anesthesiologist)
  2. Preoperative, ultrasound guided ISNB with a bupivacaine mixture: 20ml 0.5% bupivacaine and epinephrine 1:200,000.
  Arms: Standard therapy

SUMMARY:
To improve pain control and decrease opioid requirements for subjects undergoing Total Shoulder Replacement.

DETAILED DESCRIPTION:
For the pilot study the investigators will use a total of 20 cases per group.

A HIPAA Waiver will be used for screening purposes. The investigators will be using the electronic medical record system (EPIC) to screen for subjects in the University of Massachusetts Medical (UMass) system.

Subjects will be recruited and consented as described later in the study plan.

Subjects will be randomized to the two groups (standard therapy or BL) using a random number generator. The random number with the type of anesthetic will stored in envelopes and will be opened in sequence on each day of the interscalene nerve block (ISNB).

1. Group 1: Standard therapy

   1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, or age as currently determined by acute pain service (APS) anesthesiologist)
   2. Preoperative, ultrasound guided ISNB with a bupivacaine mixture: 20ml 0.5% bupivacaine and epinephrine 1:200,000.
2. Group 2: BL

   1. Standard pre-operative and post-operative medical regimen including standing acetaminophen 650mg q6hours, gabapentin 300mg q8hours and as needed oxycodone every 4 hours (unless there are contraindications due to liver function, kidney function, age, or current therapy as currently determined by APS anesthesiologist)
   2. Pre-operative ultrasound guided ISNB with a 20ml mixture consisting of 10ml of 0.5% bupivacaine with epinephrine 1:200,000, and 10ml of BL 1.33%

In accordance with our current practice, all subjects will have premedication with midazolam and fentanyl and general anesthesia (GA) with endotracheal tube (ETT). Propofol will be used for induction of GA. During surgery, administration of short acting narcotics (fentanyl) will be at the discretion of the anesthesia team.

As BL will be used, no additional local anesthetics will be used during surgery (i.e. lidocaine for induction or maintenance of anesthesia, or local anesthetics for infiltration in the surgical field). Ketamine will not be used as an anesthetic / analgesic adjunct

After this, all patients will remain on our standard protocols. In the PACU, subjects will receive IV hydromorphone for pain control. Once on the post- operative floor, subjects pain will be managed with oxycodone as needed every 4 hours (5mg for moderate pain, 10mg for severe pain) and 0.4 mg IV hydromorphone for breakthrough pain.

Subject's postoperative opioid consumption and pain scores will be obtained from their charts. Subjects will fill out a Brief Pain Inventory Short Form pre-operatively, on post-operatively day (POD) 1, and POD 2 (if the patients have not been discharged from the hospital).

Blinding In this study, the investigators will work with the Investigational Drug Pharmacy, who will store the medications, and supply medications on the day of surgery. Subjects will be blinded, as all subjects will receive an ISNB. The surgeon, anesthesiology team, post-anesthesia care unit (PACU) and floor nurses will also be unaware of group assignment, and will use their clinical judgement and subjects' reporting when administering medications and recording pain scores. Surveys about subjects' satisfaction with pain control, as well as data collection from subjects' records will be done by study investigators that are not involved in performing injections.

The Anesthesiologists performing the nerve block will not be blinded (as the Bupivacaine Liposome solution is a suspension and is white, whereas bupivacaine solution is clear), but will not participate in further evaluations of the subjects or data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects older than 18years old undergoing Total Shoulder Replacement (TSR) or reverse TSR surgery.
2. Meet criteria for regional nerve block.
3. Weight greater than 60kg (safety to keep liposomal bupivacaine and bupivacaine dosing below 3mg/kg).

Exclusion Criteria:

1. Recent drug use
2. Subjects on chronic buprenorphine therapy (either for opioid replacement or pain control).
3. Nerve injury (cervical stenosis, trauma, etc) of the surgical limb.
4. Coagulopathy
5. Subjects with significant liver disease (as amide type local anesthetics such as bupivacaine are metabolized by the liver).
6. Infection near or in the area of the nerve block.
7. Subject refusal of regional anesthesia.
8. Vulnerable populations (prisoners, mental impairment / dementia, etc).
9. Subjects requiring interpreter services (not proficient in English).
10. Subjects with poor cardio-pulmonary reserve who might not tolerate a hemi-diaphragmatic paralysis or hemi-diaphragmatic paresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Morphine Equivalent Dose of Opioids | First 24 hours
  Morphine equivalent dose (MED) of opioids within the first 24 hours after surgery (including PACU and medications on the floor)

SECONDARY OUTCOMES:
Morphine equivalent dose of opioids | 24-48 hours
  Morphine equivalent dose (MED) of opioids within the first 24-48 hours after surgery (including PACU and medications on the floor)
Visual Analogue Scale Pain Score | 24-48 hours
  Visual Analogue Scale Pain Score (VAS) in the first 24 hours, and 24-48 hours after surgery
Hospital Length of Stay | Through study completion, an average of 2-3 days
  Hospital Length of Stay
Post-Operative Brief Pain Inventory Short Form | <1 day, 1 day, and 2 days
  Brief Pain Inventory Short Form pre-operatively on POD 0, POD 1, and POD 2
Cost Analysis | Through study completion, an average of 2-3 days
  Cost estimate of each technique
Opioid Administration | Up to 72 hours
  Time to administration of the first opioid

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chan, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04134442/Prot_SAP_000.pdf